CLINICAL TRIAL: NCT02697682
Title: Treatment of Osteoarthritis With the Stromal Vascular Fraction of Abdominal Adipose Tissue - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristoffer Barfod, Consultant, MD, PHD, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OA-SVF-pilot
Record Dates: First submitted 2016-02-28; First posted 2016-03-03 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis; Stem Cells
MeSH Terms: conditions — Osteoarthritis | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): All patients are recieving the treatment.
  Interventions: Biological: injection with the stromal vascular fraction (SVF) of adipose tissue

INTERVENTIONS:
Biological: injection with the stromal vascular fraction (SVF) of adipose tissue — Description of the active treatment The active treatment is an intra-articular injection with the stromal vascular fraction (SVF) harvested from the patient's own abdominal subcutaneous fatty tissue. SVF is harvested using the Lipogems system.

SUMMARY:
To investigate the feasibility and short term safety issues of treatment of knee osteoarthritis with intra-articular injection with the stromal vascular fraction of abdominal adipose tissue (SVF) harvested and prepared using the Lipogems System.

Hereby we wish to pave the road for a high quality randomized controlled trial investigating effectiveness of treatment of knee osteoarthritis with SVF looking at patient reported outcome, function, homeostasis of the joint and cartilage regeneration.

DETAILED DESCRIPTION:
Background Osteoarthritis (OA) of the knee is a destructive joint disease, causing degeneration of cartilage, damage to the underlying bone and morphological changes to the joint1. It is a major public health concern due to the increased life expectancy of the ageing population2,3. No approved medical treatment that reverses the morphological changes currently exists. Conventional treatment includes physiotherapy, pain killers, braces and in end-stage OA surgical knee replacement4.

Treatment of Osteoarthritis with Paqe 3 Version 2 the Stromal Vascular Fraction of Adipose tissue 02-11-2015 During the past decade researchers have started to explore the regenerative potential of mesenchymal stem cells (MSC) in OA5. MSCs are multipotent progenitor cells able to give rise to osteocytes, adipocytes, chondrocytes, myoblasts and tenocytes6. MSCs were first used to treat Chondral defects in 19987 and to treat OA in 20028. Since, a number of case reports and prospective series have been published showing significant short term and long term effect on pain and cartilage thickness5. Recently a prospective case-series of 1128 patients involving 1856 joints were treated with the stromal vascular fraction of abdominal Adipose tissue (SVF) which is a rich source of mesenchymal stem cells. 86% of the treated patients showed an improvement of at least 50% in modified Knee/Hip Osteoarthritis Outcome Score (KOOS/HOOS) at 3 months and 129. Only 0.9% of patients were non-responders showing no improvement after treatment. No serious adverse effects like infection or tumor formation were observed9, which is in accordance with previous studies10. Non-manipulated or minimally manipulated cell therapies have been used within a wide range of medical conditions including: stroke, myocardial infarction, Crohn's disease, rheumatoid arthritis and breast augmentation. More than 17,000 scientific articles have been published reporting treatment of more than 320,000 patients11. No severe safety issues have been raised12.

Mesenchymal stem cells can be derived from bone marrow or adipose tissue5. Most research has been performed on bone marrow-derived stem cells but the past years a series of studies have been published showing promising effect of Adipose-derived mesenchymal stem cells (AMSCs). By using AMSC a large amount of cells can be harvested from a small volume of tissue thereby avoiding the costly and time consuming process of expanding the cells in culture5,9. Abdominal adipose tissue has been shown to have a 1000 times higher concentration of AMSC than other investigated adipose tissue9. This opens for the possibility of a one-step procedure where cells are harvested and injected during one visit in the outpatient clinic. The optimal dose of AMSC is unknown but the effect seems to be dose-dependent with doses around 1.0 x 108 AMSCs per injection being desirable5,9. The stromal vascular fraction of abdominal Adipose tissue is a rich source of adipose derived mesenchymal stem cells.

In 2014 the Lipogems system has been launched as a commercial of-the-shelf product: http://lipogems.eu/. The Lipogems system is an enzyme-free technology developed to process lipoaspirates in a closed system, resulting in a non-expanded adipose tissue product that contains SVF13. Before using this product in larger scale a controlled study of its feasibility and safety is needed.

Study Objective To investigate the feasibility and short term safety issues of treatment of knee osteoarthritis with intra-articular injection with the stromal vascular fraction of abdominal adipose tissue (SVF) harvested and prepared using the Lipogems System.

Hereby we wish to pave the road for a high quality randomized controlled trial investigating effectiveness of treatment of knee osteoarthritis with SVF looking at patient reported outcome, function, homeostasis of the joint and cartilage regeneration.

6 Treatment Patients participating in the study are treated according to the Danish National Clinical Guidelines for people with osteoarthritis16. They receive three months of physiotherapy, are guided concerning the optimal pharmaceutical treatment with painkillers and people with BMI above 28 are offered a consultation with a dietitian.

6.1 Description of the active treatment The active treatment is an intra-articular injection with the stromal vascular fraction (SVF) harvested from the patient's own abdominal subcutaneous fatty tissue. SVF is harvested using the Lipogems system.

6.1.1 Harvest of SVF Harvest of SVF is done under sterile conditions in the outpatient clinic. The patient is positioned supine on an examination bench. The area from which the tissue will be harvested is marked on the skin with a surgical marker. The area is app. 8cm (cranio-caudal) x 20cm (lateral) and situated just below the umbilicus. Local anesthesia is applied to the whole area with a suspension of Carbocain 1%, 200ml isotonic saline, adrenaline and 10mmol Bicarbonate. Surgical cleaning is performed twice and a sterile draping is applied. Through a stab incision the harvesting needle is introduced to the subcutaneous fat and suction is applied. 20ml to 40ml of subcutaneous adipose tissue is harvested. At the end of the procedure the skin is closed with a plaster.

6.1.2 Preparation of SVF for implantation The syringes with subcutaneous aspirate are prepared using the Lipogems system. The Lipogems system is an enzyme-free technology developed to process variable amounts of lipoaspirates in a closed system, resulting in a nonexpanded adipose tissue product that contains SVF. The technology works through a mild mechanical tissue cluster size reduction. Thereby avoiding the use of any enzyme and additional processing (i.e., centrifugation and subfractional harvesting).13 6.1.3 Implantation of SVF Implantation of the SVF is done under sterile conditions in the outpatient clinic. The patient is positioned supine on an examination bench with the affected knee stretched. The superior pole of the patella is palpated and the femoral condyle is marked with a surgical marker. The suprapattelar recess is located by ultrasound, local anesthesia is applied to the injection site and surgical cleaning is performed twice. Injection of the SVF in to the suprapattelar recess is done using a 21 gauge syringe under direct visualization by ultrasound. At the end of the procedure the skin is closed with a plaster.

6.1.4 Control of dose of injected SVF Control of the dose of AMSC in the injected SVF is performed after injection. As a consequence of the logistical favorable setup where harvest and implantation is performed in a one-step procedure it is not possible to count the AMSC before injection. Instead one mL of the solution is sent for cell count in the pathological department.

ELIGIBILITY:
Inclusion Criteria:

Age 18-70 years. Kellgren-Lawrence grade 1 - 4 evaluated on x-ray or ICRS grade 2-4 evaluated on MRI.

The patient must be expected to be able to attend rehabilitation and post-examinations.

The patient must be able to speak and understand Danish. The patient must be able to give informed consent.

Exclusion Criteria:

Varus or valgus malalignment of the knee > 5 degrees. BMI > 35 Terminal illness or severe medical illness: ASA score higher than or equal to 3.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | 3 months
  An adverse event is defined as any event caused by the treatment leading to a less preferable situation for the patient. Patients will be screened for:
  Donor site morbidity: (Infection, swelling, pain). Implant site morbidity: (Infection, swelling, pain (increased VAS score))

SECONDARY OUTCOMES:
The Knee injury and Osteoarthritis Outcome Score | 3+12 months
  The KOOS holds 42 items in five separately scored subscales: KOOS Pain, KOOS Symptoms, Function in daily living (KOOS ADL), Function in Sport and Recreation (KOOS Sport/Rec), and knee-related Quality of Life (KOOS QOL)
Numeric Rating Scale for Assessment of Pain Intensity | 3+12 months
  For assessment of pain intensity, the 11-step numeric rating scale (NRS-11) is chosen. The scale goes from 0 to10, with 0 equalling no pain and 10 being the worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Barfod, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital Koege, Koege, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barfod KW, Blond L. Treatment of osteoarthritis with autologous and microfragmented adipose tissue. Dan Med J. 2019 Oct;66(10):A5565. PMID 31571571